CLINICAL TRIAL: NCT02259569
Title: Comparison of Peak Airway Pressure and Gastric Insufflation in Pressure-Controlled Ventilation or Volume-Controlled Ventilation With I-Gel in Pediatric Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2014-0594
Record Dates: First submitted 2014-09-22; First posted 2014-10-08 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Pediatric Urologic Surgeries
Keywords: Gastric insufflation; I-gel; Peak airway pressure; Pressure-controlled ventilation; Volume-Controlled Ventilation; pediatric patient

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCV group (Experimental): After insertion of I-gel, mechanical ventilation of the lungs was commenced. Mechanical ventilator was set to obtain a tidal volume of 8ml/kg in pressure-controlled mode.
  Interventions: Other: Pressure-controlled ventilation
- VCV group (Active Comparator): After insertion of I-gel, mechanical ventilation of the lungs was commenced. Mechanical ventilator was set to obtain a tidal volume of 8ml/kg in volume-controlled mode.
  Interventions: Other: Volume-controlled ventilation

INTERVENTIONS:
Other: Pressure-controlled ventilation
  Arms: PCV group
Other: Volume-controlled ventilation
  Arms: VCV group

SUMMARY:
The purpose of this study is to compare peak airway pressure and gastric insufflation in Pressure-Controlled Ventilation or Volume-Controlled Ventilation with I-Gel in pediatric patient

ELIGIBILITY:
Inclusion Criteria:

① ASA I-II patients aged between 1 and 7 year undergoing elective urologic surgery.

Exclusion Criteria:

* parent refusal

  * clinically significant respiratory disease ③ congenital airway abnormalities, oropharyngeal or facial pathology ④ risk of aspiration

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Gastric insufflation determined by increase of cross sectional area of gastric antrum, measured by ultrasonography. | 1 min after I-gel insertion

SECONDARY OUTCOMES:
oropharyngeal leak pressure | 1 min after caudal block
FOB grade | 1 min after I-gel insertion
  grade 1= only the vocal cords visible, 2= vocal cords and epiglottis visible, 3= only the epiglottis visible, 4= vocal cords and epiglottis not visible
peak airway pressure | 1 min after I-gel insertion

OTHER OUTCOMES:
dynamic compliance | 1 min after end of surgery
typical gurgle or whoosh sound | 1 min after caudal block
  gastric insufflation determined by continuous epigastric auscultation